CLINICAL TRIAL: NCT02256956
Title: Effects of Amitriptyline on Central Pain Processing in Healthy Volunteers Depending on CYP Pharmacogenetics
Brief Title: Genetic Determinants of Amitriptyline Efficiency for Pain Treatment - Part II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Washington (Other); Aalborg University (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 133/12_2
Record Dates: First submitted 2014-09-29; First posted 2014-10-06 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pain
Keywords: Pharmacogenetics of Amitriptyline
MeSH Terms: conditions — Chronic Pain | interventions — Amitriptyline; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amitriptyline first, Placebo second (Active Comparator): Amitriptyline first, Placebo second
  Interventions: Drug: Amitriptyline; Drug: Tolterodine
- Placebo first, Amitriptyline second (Active Comparator): Placebo first, Amitriptyline second
  Interventions: Drug: Amitriptyline; Drug: Tolterodine

INTERVENTIONS:
Drug: Amitriptyline — 25 mg / day for 10 days
  Other Names: Tryptizol
Drug: Tolterodine — Placebo 1 mg / day for 10 days

SUMMARY:
Low dose tricyclic antidepressant drugs are routinely administered co-analgesics in pain medicine. Amitriptyline is largely considered as a gold standard. Amitriptyline underlies cytochrome CYP2D6 and CYP2D19 metabolism. CYP2D6 is highly polymorphic; numerous genetic variants result in 4 major classes characterizing enzymatic activity: poor metabolizers, intermediate metabolizers, extensive metabolizers and ultrarapid metabolizers. It is not known to which extent metabolizer classes determine pain outcomes or side-effects. As only one in three pain patients is considered to be a responder to amitriptyline's co-analgesic effect, prediction of treatment efficacy with a fast and easy to perform bedside test may contribute to the patients quality of life. The aim of this study is to determine the influence of cytochrome variants on experimental pain, drug related side-effects and finally identification of active metabolites.

DETAILED DESCRIPTION:
Background

Pain is defined as an ongoing unpleasant sensory experience, which can be classified according to three major, although overlapping, etiologies: nociceptive, inflammatory and neuropathic pain.

Antidepressants are widely used as co-analgesics in the management of chronic pain. An overview of different substances and their relation to their mechanism of action is presented in the review of Dharmashaktu et al. Low-dose tricyclic antidepressants are well established in the treatment of neuropathic pain. Amitriptyline and imipramine are two widely used substances of this group. The hypoalgesic effect of amitriptyline is mainly mediated by inhibiting serotoninergic and noradrenergic reuptake. When administered at night time, amitriptyline's sedating effect enhances sleep quality, considered as an important improvement in quality of life in chronic pain patients.

Tricyclic antidepressants undergo biotransformation in the liver with CYP2D6 catalyzing hydroxylation, whereas CYP2C19 mediates demethylation of the parent drug. The demethylated metabolites are partially tricyclic drugs by themselves, such as nortriptyline and desipramine, which are demethyl-metabolites of amitriptyline and imipramine. It is unknown whether the analgesic effect of amitriptyline is mediated through its precursor or the metabolites.

The CYP2D6 gene is highly polymorphic and the numerous genetic variants result in 4 major metabolizer classes characterizing enzyme activity: poor metabolizers (PM) with no enzyme activity, intermediate metabolizers (IM) with reduced enzyme activity, (EM) extensive metabolizers carrying two functionally active alleles and ultrarapid metabolizers (UM) carrying a gene duplication or multi-duplication resulting in increased enzyme activity.

CYP2D6 PMs have higher plasma concentrations of the parent drug than EMs and are, therefore, more likely to experience dose-dependent adverse drug reactions. In 50 psychiatric patients receiving amitriptyline 150 mg/d, carriers of two functional CYP2D6 alleles (EMs) had a significantly lower risk of side effects than IM (12.1% vs. 76.5%). The lowest risk was observed for carriers of two functional CYP2D6 alleles combined with only one functional CYP2C19 allele. The combination of normal (fast) CYP2C19 and slightly diminished CYP2D6 function leads to high concentrations of toxic intermediate metabolites and an increase of adverse events. On the other hand, CYP2D6 UMs may be at risk for sub-therapeutic concentrations resulting in poor therapeutic response. Thus, genetically determined differences in blood concentrations of antidepressants make dose adjustments advisable. However, these findings and dose recommendations have only been evaluated for psychiatric patients and no investigation on antidepressants as low-dosed co-analgesics are available up to now.

Quantitative sensory tests (QST) have been intensively used for more than three decades to explore the central processing of painful stimuli in patients and healthy volunteers. QST were developed to assess the responses to sensory stimuli, providing psychophysical methods for the assessment of the nociceptive system. In addition, large cohorts of healthy volunteers have been investigated using QST measures to produce reference values.

QST measures are based on a multimodal and multi-tissue approach, combining different pain modalities applied to different tissues in order to gather sufficient and discriminative information about the human nociceptive system. QST will be our tool to characterize analgesic efficacy of amitriptyline. QST offers the unique opportunity of experimentally induced pain being quantitatively measured by psychophysical, behavioural and neurophysiological responses.

Objective

We test the hypothesis that the extensive and ultrarapid CYP2D6 metabolizers are associated with a higher analgesic effect of amitriptyline, compared to the poor and intermediate metabolizers, as assessed by quantitative sensory tests. Plasma concentrations of amitriptyline and its metabolites will be analysed as co-variates for drug efficacy.

Two sub-studies, one peak-level, single-dose administration and one steady-state, repeated dose administration, are needed to assess the pharmacokinetics of amitriptyline and its active metabolites.

Statistics are provided by José A. Biurrun Manresa.

Methods

Two consecutive randomized placebo-controlled two-way crossover sub-studies on amitriptyline will be conducted in consenting, healthy, male volunteers. Both sub-studies have the same aim: to determine the association between CYP2D6 genotype, drug response measured by QST and plasma concentrations of amitriptyline and its metabolites. The first sub-study will be conducted with a single high dose of amitriptyline (100 mg). This sub-study will be conducted with repeated low doses of amitriptyline (25 mg) once a day for 10 days.

In both sub-studies the same experimental procedures and statistical analyses will be performed. The only difference between the sub-studies is the dose of amitriptyline and the duration of drug intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* >7 Metabolic Equivalents
* Written informed consent

Exclusion Criteria

* Chronic pain syndrome
* Drug abuse
* Alcohol abuse
* Suspicion of neurologic dysfunction at tested sites
* Ongoing treatment with antidepressants
* Ongoing treatment with analgesics
* Pretreatment with any CYP3A inducers or inhibitors
* Known allergy to tested drugs
* Elevated eye pressure
* Obstructive uropathy
* Heart disease
* Pulmonary disease
* Neurological disease
* Psychiatric illness

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2018-05 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Nociceptive withdrawal reflex | During measurement, expected to be ca. 2-3 minutes
  Measure of involuntary electromyographic amplitude

SECONDARY OUTCOMES:
Pharmacogenetic information on CYP2D6 metabolism | At baseline, i.e. on day 1
  Laboratory measurement (genotyping)
Changes in plasmatic metabolite level | Throughout study duration, expected to be ca. 20 days
  Metabolite level in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Stamer, Professor, Study Chair — Bern University Hospital; Pascal H Vuilleumier, MD, Principal Investigator — Bern University Hospital
Locations (1):
- Dep. of Anesthesiology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Dharmshaktu P, Tayal V, Kalra BS. Efficacy of antidepressants as analgesics: a review. J Clin Pharmacol. 2012 Jan;52(1):6-17. doi: 10.1177/0091270010394852. Epub 2011 Mar 17. PMID 21415285